CLINICAL TRIAL: NCT02333864
Title: POGO® Automatic Blood Glucose Monitoring System Clinical Study
Status: Completed | Type: Observational
Sponsor: Intuity Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-000321
Record Dates: First submitted 2014-12-17; First posted 2015-01-07 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PWD testing POGO® BGMS: All enrolled persons with diabetes
  Interventions: Device: POGO® BGMS

INTERVENTIONS:
Device: POGO® BGMS — SMBG

SUMMARY:
The purpose of this study is to determine if the POGO® system delivers accurate blood glucose readings in the hands of the lay user and assess the POGO® system accuracy when used by trained health care professionals.

DETAILED DESCRIPTION:
Subjects will review labeling materials and self-test using the POGO® system. An HCP-assisted test also will be performed; both tests will be compared to a fingerstick capillary sample run on a YSI reference glucose analyzer. Subjects will complete questionnaires on labeling comprehension and POGO® usability.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with diabetes
* Be 18 years of age or older
* Be able to read, write, and understand English fluently
* Be able and willing to give written informed consent and have provided signed, written consent

Exclusion Criteria:

* Any condition which in the opinion of the Investigator may place the subject or site personnel at excessive risk
* A physical condition or limitation that prevents the subject from reading the labeling and using a BGMS on their own
* Previous experience with the POGO® BGMS
* Formal experience with clinical (medical) laboratory equipment or formal training in a relevant medical field

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who are 18 years of age or older and have been diagnosed with diabetes
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Accuracy Validation of the POGO® BGMS: Minimum outcome of 95% of results within 20% of reference measurement. | Blood glucose measured at time of single visit for each subject, endpoint evaluated at completion of study (approximately four months after initiation.)
  Lay-user accuracy
Accuracy Verification of the POGO® BGMS: Minimum outcome of 95% of results within 20% of reference measurement. | Blood glucose measured at time of single visit for each subject, endpoint evaluated at completion of study (approximately four months after initiation.)
  HCP accuracy

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Diablo Clinical Reasearch, Walnut Creek, California
  - Park Nicollett Institute - International Diabetes Center, Minneapolis, Minnesota